CLINICAL TRIAL: NCT02034539
Title: Prospektive, Randomisierte Und Kontrollierte Studie Zum Einfluss Des VADOplex-Systems Auf Die Lebensqualität im Rahmen Der Behandlung Der Chronisch-kritischen Extremitätenischämie im Stadium IV Nach Fontaine
Brief Title: VADOplex Critical Limb Ischemia Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Collaborators: OPED GmbH (Unknown)
Responsible Party: Principal Investigator, Claas Luedemann, Claas Luedemann, MD, Asklepios Kliniken Hamburg GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VADOplex-1
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Peripheral Artery Disease; Quality of Life; Wound Healing
Keywords: peripheral artery disease; critical limb ischemia; VADOplex; intermittent foot compression
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VADOplex treatment (Experimental): best medical treatment in combination with intermittent pneumatic foot compression by the VADOplex system for 4 - 6 hours/day until total wound closure of the target lesion is achieved with a maximum treatment of 24 weeks
  Interventions: Device: VADOplex system
- conservative treatment (No Intervention): best medical treatment of the target lesion alone

INTERVENTIONS:
Device: VADOplex system — intermittent automatic pneumatic compression of the sole of the foot by the VADOplex system
  Arms: VADOplex treatment

SUMMARY:
In patients with critical limb ischemia (CLI) and foot ulcers wound healing is an important goal which can normally only be achieved after sufficient treatment of the underlying ischemia (revascularization either by an operation, e. g. bypass, or a catheter intervention). After successful revascularization everything should be done to improve wound healing because this regularly takes weeks up to several months. One possibility to speed up healing could be treatment with the VADOplex device which delivers an automatic intermittent painless compression of the sole of the foot thereby increasing perfusion of the leg. This system can be easily operated by patients themselves and at home.

Our goal is to prove that the VADOPlex system accelerates healing up and improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

* signed informend consent
* peripheral artery disease Fontaine IV (equals Ruterford 5 and 6) with or without neuropathy
* foot lesion stage 1 - 4 analogous to 4 Wagner classification of the diabetic foot
* secondary wound healing if previous surgical wound treatment
* previous interventional and/or surgical revascularisation
* age above 18
* hosptalized to the beginning of the study

Exclusion Criteria:

* primary wound healing if previous surgical wound treatment
* uncontrolled local or systemic infection
* renal failure on dialysis
* inability or insufficient help to operate the VADOplex system
* wound dressings that lead to insufficient compression by the VADOplex system (e.g. total contact cast for offloading)
* wounds of other than ischemic or neuro-ischemic origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
wound healing | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  complete healing of the target lesion
change of quality of life | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  change of quality of life compared to baseline. Quality of life measured with the EQ-5D tool (European quality of life in 5 dimensions)

SECONDARY OUTCOMES:
time to complete wound healing | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  time until complete wound healing of the target lesion is achieved
Wound size | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  overall reduction of the size of the target lesion in patients with incomplete wound healing compared to baseline
change of pain intensity | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  change of pain intensity compared to baseline. Pain intensity measured with a numeric rating scale (0 - 10) or if not applicable with a visual analogue scale
change of ankle-brachial index | at discharge, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 24 weeks after discharge
  change of ankle-brachial index compared to basleline
incidence of deep vein thrombosis | 24 weeks after discharge or whenever a thrombosis is suspected

CONTACTS AND LOCATIONS:
Overall Officials: Holger Lawall, MD, Principal Investigator — head of department
Locations (1):
- Gefäßzentrum, Asklepios Westklinikum Hamburg, Hamburg, Hamburg, Germany